CLINICAL TRIAL: NCT04313010
Title: Effectiveness of Regenerative Endodontics Therapy for Single-rooted Mature Permanent Tooth With Pulp Necrosis: a Multicenter Randomized Controlled Clinical Trial.
Brief Title: Effectiveness of Regenerative Endodontics Therapy for Single-rooted Mature Permanent Tooth With Pulp Necrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Collaborators: Shenzhen Hospital, Southern Medical University (Unknown)
Responsible Party: Principal Investigator, Wanghong Zhao, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC2019ZD023
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pulp Necrosis
Keywords: Pulp Necrosis; Regenerative Endodontics Therapy; Platelet Rich Fibrin
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regenerative endodontics therapy with PRF (Experimental): In the procedures of regenerative endodontics therapy, K-files were intentionally used to violate the periapical tissues via overinstrumentation up to 2-3mm past the apical foramen to induce bleeding. Only the apex 1/3 of the root canal need to be filled with blood. PRF was injected into the root canal to a level below the CEJ, then wait for 10-15min to coagulate.
  Interventions: Other: PRF
- Regenerative endodontics therapy with BC (Active Comparator): In the procedures of regenerative endodontics therapy, K-files were intentionally used to violate the periapical tissues via overinstrumentation up to 2-3mm past the apical foramen to induce bleeding. The adequate blood need to be full with canal space and below the CEJ, then wait for 10-15min to coagulate.
  Interventions: Other: BC

INTERVENTIONS:
Other: PRF — A sample of whole venous blood was drawn from the patient's forearm. The blood sample was transferred into a tube without anticoagulant and centrifuged immediately using a centrifuge.
  Arms: Regenerative endodontics therapy with PRF
Other: BC — According to the procedures of regenerative endodontics therapy, BC was made by the way of provoking apical bleeding into root canal.
  Arms: Regenerative endodontics therapy with BC

SUMMARY:
This study is to evaluate the effectiveness of regenerative endodontics therapy in single-rooted permanent teeth with pulp necrosis，and compare the clinical efficacy of platelet rich fibrin (PRF) and blood clot (BC) as scaffolds.

DETAILED DESCRIPTION:
Regenerative endodontics therapy (RET), based on the principles of tissue engineering, manipulates stem cells, scaffold, and bioactive growth factors to achieve the functional reconstruction of pulp tissue. RET has been recommended strongly as an alternative in treating immature permanent teeth with necrotic pulp in recent years, while root canal therapy (RCT) has been extensively applied in the treatment of mature permanent teeth with necrotic pulp. RCT contains the chemomechanical preparation of the infected root canals to eliminate the microorganisms, and root canal obturation with filling materials to reduce and prevent microbial contamination in root canal system. However, the root canal filling materials, such as Gutta-percha, are inert materials which fail to recover the physiological function of the pulp. As RET has been proved curative for immature permanent teeth diagnosed with pulp necrosis, doctors and researchers try to extend its application in the mature ones. Encouragingly, several RET cases for mature teeth reported in the literature have shown positive clinical outcomes. However, it still lacks long-term and well-designed randomized clinical trial with large sample size and following standardized protocol, hence this study is conducted to make up for it to achieve high-level evidence.

In the process of RET, the scaffold can provide nutrition and space, which are essential for the proliferation and differentiation of stem cells. Therefore, it is a crucial step to select a high-quality material as the scaffold. In many studies of RET procedures, blood clot (BC), generated by provoking apical bleeding into the root canal, is regarded as a scaffold. Nevertheless, it remains a common problem that operators may fail to induce apical bleeding or achieve adequate blood volume. Recent studies suggest that patelet rich fibrin (PRF), the second-generation platelet concentrate, can provide a fibrin network full of cytokines and growth factors, which may improve the desired biological outcome. Accordingly, we assumed that PRF could improve the curative effect for mature teeth in RET. The purpose of this study is to compare the clinical efficacy of PRF and BC as scaffolds in RET for the mature permanent tooth with pulp necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Intended to participate with this study, and provide informed assent/consent.
* Aged 10 and 59 years.
* At least one mature permanent teeth diagnosed as pulp necrosis with or without periapical lesion, and CBCT showed the teeth has single root and single root canal.

Exclusion Criteria:

* Allergic to any medications or materials necessary to complete the procedures.
* The teeth with severe coronal defect, of which pulp space is needed for post/core final restoration.
* Non-restorable teeth.
* The teeth with root fracture or vertical root fractures.
* Concurrent signs of other pathological root resorption.
* Patients with periodontitis.
* Patients with dental dysplasia or other oral genetic disorders.
* Women who are pregnant or lactating, or women who plan to become pregnant in the subsequent 2 years.
* Patients with dental phobia.
* Patients with mental disorders.
* Patients with a history of systemic diseases that may alter immune function.
* Patients with medical conditions and/or receiving medications that would affect patients' body's ability of healing or blood clotting.
* Participants who are participating in or had participated in other clinical studies within the prior 3 months.

Ages: 10 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 346 (Estimated)
Dates: Start 2020-03-16 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Success of regenerative endodontics therapy | 24 months
  Success: Defined as symptoms, clinical and radiographic assessment of the teeth. The teeth with RET were asymptomatic; Clinical examination showed absence of clinical signs of pain and soft tissue pathology (e.g. abscess, sinus tract etc.). Radiographic assessment showed the reduction and/or absence of periapical radiolucency.

SECONDARY OUTCOMES:
Change in pulp vitality | 1、3、6、12、18、24 months
  Change in pulpal vitality will be assessed through pulpal response to sensitivity tests (cold, hot and electrical test) in teeth treated with RET.
Adverse events | 1、3、6、12、18、24 months
  Such as discoloration, reinfection, root resorption and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Wanghong Zhao, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (3):
- China (3):
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Stomatological Hospital, Southern Medical University, Guangzhou
  - Shenzhen Hospital, Southern Medical University, Shenzhen

REFERENCES:
- [Background] Kim SG, Malek M, Sigurdsson A, Lin LM, Kahler B. Regenerative endodontics: a comprehensive review. Int Endod J. 2018 Dec;51(12):1367-1388. doi: 10.1111/iej.12954. Epub 2018 Jun 11. PMID 29777616
- [Background] Diogenes A, Ruparel NB, Shiloah Y, Hargreaves KM. Regenerative endodontics: A way forward. J Am Dent Assoc. 2016 May;147(5):372-80. doi: 10.1016/j.adaj.2016.01.009. Epub 2016 Mar 24. PMID 27017182
- [Background] Adnan S, Ullah R. Top-cited Articles in Regenerative Endodontics: A Bibliometric Analysis. J Endod. 2018 Nov;44(11):1650-1664. doi: 10.1016/j.joen.2018.07.015. Epub 2018 Sep 19. PMID 30243658
- [Background] Saoud TM, Sigurdsson A, Rosenberg PA, Lin LM, Ricucci D. Treatment of a large cystlike inflammatory periapical lesion associated with mature necrotic teeth using regenerative endodontic therapy. J Endod. 2014 Dec;40(12):2081-6. doi: 10.1016/j.joen.2014.07.027. Epub 2014 Oct 5. PMID 25292168
- [Background] Saoud TM, Martin G, Chen YH, Chen KL, Chen CA, Songtrakul K, Malek M, Sigurdsson A, Lin LM. Treatment of Mature Permanent Teeth with Necrotic Pulps and Apical Periodontitis Using Regenerative Endodontic Procedures: A Case Series. J Endod. 2016 Jan;42(1):57-65. doi: 10.1016/j.joen.2015.09.015. Epub 2015 Oct 31. PMID 26525552
- [Background] Paryani K, Kim SG. Regenerative endodontic treatment of permanent teeth after completion of root development: a report of 2 cases. J Endod. 2013 Jul;39(7):929-34. doi: 10.1016/j.joen.2013.04.029. Epub 2013 May 14. PMID 23791266
- [Background] Nageh M, Ahmed GM, El-Baz AA. Assessment of Regaining Pulp Sensibility in Mature Necrotic Teeth Using a Modified Revascularization Technique with Platelet-rich Fibrin: A Clinical Study. J Endod. 2018 Oct;44(10):1526-1533. doi: 10.1016/j.joen.2018.06.014. Epub 2018 Aug 31. PMID 30174103
- [Background] Galler KM, Krastl G, Simon S, Van Gorp G, Meschi N, Vahedi B, Lambrechts P. European Society of Endodontology position statement: Revitalization procedures. Int Endod J. 2016 Aug;49(8):717-23. doi: 10.1111/iej.12629. Epub 2016 Apr 23. PMID 26990236
- [Background] Ulusoy AT, Turedi I, Cimen M, Cehreli ZC. Evaluation of Blood Clot, Platelet-rich Plasma, Platelet-rich Fibrin, and Platelet Pellet as Scaffolds in Regenerative Endodontic Treatment: A Prospective Randomized Trial. J Endod. 2019 May;45(5):560-566. doi: 10.1016/j.joen.2019.02.002. Epub 2019 Mar 30. PMID 30935618
- [Background] Varela HA, Souza JCM, Nascimento RM, Araujo RF Jr, Vasconcelos RC, Cavalcante RS, Guedes PM, Araujo AA. Injectable platelet rich fibrin: cell content, morphological, and protein characterization. Clin Oral Investig. 2019 Mar;23(3):1309-1318. doi: 10.1007/s00784-018-2555-2. Epub 2018 Jul 12. PMID 30003342
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Derived] Liang Y, Ma R, Chen L, Dai X, Zuo S, Jiang W, Hu N, Deng Z, Zhao W. Efficacy of i-PRF in regenerative endodontics therapy for mature permanent teeth with pulp necrosis: study protocol for a multicentre randomised controlled trial. Trials. 2021 Jul 6;22(1):436. doi: 10.1186/s13063-021-05401-7. PMID 34229752